CLINICAL TRIAL: NCT03969329
Title: Phase 3, Single-arm, Open-label, Multidose, Titration, Pharmacokinetic, Pharmacodynamic, and Safety Study of Etelcalcetide in Children and Adolescents ≥ 2 to < 18 Years of Age With Secondary Hyperparathyroidism and Chronic Kidney Disease Receiving Maintenance Hemodialysis
Brief Title: A Phase 3 Study of Etelcalcetide in Children With Secondary Hyperparathyroidism Receiving Hemodialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170724
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary hyperparathyroidism (sHPT); Chronic kidney disease (CKD); Paediatric
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Intervention Model Description: Participants will remain on treatment for 26 weeks from day 1 or until the time of renal transplant or parathyroidectomy, whichever occurs first. Participants will receive a starting dose of etelcalcetide 0.07 mg/kg or 5 mg, whichever is lower, 3 times a week (TIW) intravenously. The dose of etelcalcetide will be titrated every 4 weeks (weeks 5, 9, 13, and 17) based on intact parathyroid hormone (iPTH), calcium, and safety to a maximum dose of 0.21 mg/kg or 15 mg, whichever is lower. The lowest protocol specified dose (PSD) for this trial is 0.035 mg/kg or 2.5 mg, whichever is lower.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Etelcalcetide (Experimental): Participants will receive etelcalcetide in addition to standard of care.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Etelcalcetide has been shown to be safe and efficacious in treating adult CKD patients with SHPT by simultaneously controlling iPTH, calcium (Ca), and phosphorus and has recently been approved for use in adult patients with SHPT treated with hemodialysis in both the United States and Europe.
  Other Names: Parsabiv - brand name

SUMMARY:
Assess the efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of etelcalcetide in the treatment of secondary hyperparathyroidism (SHPT) in pediatric participants between ≥ 2 to < 18 years of age, with chronic kidney disease (CKD) on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant's legally acceptable representative has provided informed consent when the participant is legally too young to provide informed consent and the participant has provided written assent based on local regulations and/or guidelines prior to any trial-specific activities/procedures being initiated.
* Male or female participants greater than or equal to 2 to less than 18 years of age at the time of enrollment.
* Targeted dry weight greater than or equal to 7 kg at the time of screening Week -1.
* Diagnosed with CKD and SHPT undergoing hemodialysis/hemodiafiltration TIW or four times a week (QIW) at the time of screening greater than or equal to 1 month.
* Diagnosis of SHPT with the mean of the 2 consecutive central laboratory iPTH values greater than 300 pg/mL during screening, on separate days and within 2 weeks of enrollment obtained from the central laboratory during screening.
* Serum corrected Ca value greater than or equal to 9.0 mg/dL obtained from the central laboratory during screening.
* Dialysate Ca level greater than or equal to 2.5 mEq/L for at least 1 month prior to screening and throughout the duration of the trial.
* participant receiving active vitamin D sterols must have had no more than a maximum dose change of 50% within the 2 weeks prior to screening laboratory assessments, remain stable through enrollment, and be expected to maintain stable doses for the duration of the trial, except for adjustments allowed per protocol.
* participant receiving phosphate binders must have had no more than a maximum dose change of 50% within the 2 weeks prior to screening laboratory assessments, remain stable through enrollment, and be expected to maintain stable dose for the duration of the trial, except for adjustments allowed per protocol.
* Subject receiving Ca supplements must have had no more than a maximum dose change of 50% within the 2 weeks prior to screening laboratory assessments, remain stable through enrollment, and be expected to maintain stable dose for the duration of the trial, except for adjustments allowed per protocol.
* SHPT not due to vitamin D deficiency, per investigator assessment.

Exclusion Criteria:

* Disease Related:
* History of congenital long QT syndrome, second or third degree heart block, ventricular tachyarrhythmia's, history of symptomatic ventricular dysrhythmias Torsades de Pointes or other conditions associated with prolonged QT interval.
* Anticipated or scheduled parathyroidectomy during the trial period.
* Anticipated or scheduled kidney transplant during the trial period.
* Participant has received a parathyroidectomy within 6 months prior to enrollment.
* Other Medical Conditions:
* Current malignancy or history of other malignancy, except non-melanoma skin cancers within the last 5 years.
* Prior/Concomitant Therapy:
* Use of concomitant medications that may prolong the QTc (eg, ondansetron, albuterol, sotalol, amiodarone, erythromycin, or clarithromycin). Refer to CredibleMeds.org for guidance. Certain medications may be allowed based on review by the Medical Monitor and require additional electrocardiogram (ECG) monitoring and potential electrolyte monitoring.
* Receipt of cinacalcet therapy within 30 days prior to screening and through enrollment.
* Any previous use of etelcalcetide prior to screening and through enrollment (Original protocol, Amendment 1, and Amendment 2 only).
* Receipt of etelcalcetide therapy within 6 months prior to screening assessments and through enrollment (Amendment 3 and later only).
* All herbal medicines (eg, St. John's wort), vitamins, and supplements consumed by the participant within the 30 days prior to enrollment, and continuing use if applicable, will be reviewed by the Principal Investigator and the Amgen Medical Monitor. Written documentation of the review and Amgen acknowledgment is required for participant participation.
* Use of any over-the-counter or prescription medications within the 14 days or 5 half-lives (whichever is longer) prior to enrollment that are not established therapies for participants with renal disease or other conditions secondary to renal disease will be reviewed by the Principal Investigator and the Amgen Medical Monitor. Written documentation of the review and Amgen acknowledgment is required for participant participation. Paracetamol for analgesia will be allowed.
* Prior/Concurrent Clinical Trial Experience:
* Currently receiving treatment in another investigational device or drug trial, or less than 30 days since ending treatment on another investigational device or drug trial(s). Other investigational procedures while participating in this trial are excluded.
* Diagnostic Assessments During Screening:
* Participant has significant abnormalities on the most recent central laboratory test during the screening period prior to enrollment per the Investigator including but not limited to the following: a. Serum transaminase (alanine aminotransferase [ALT] or serum glutamic pyruvic transaminase [SGPT], aspartate aminotransferase [AST], or serum glutamic oxaloacetic transaminase [SGOT]) greater than 1.5 times the upper limit of normal (ULN).
* Corrected QT interval greater than 500 ms, using Bazett's formula.
* Corrected QT interval greater than or equal to 450 to less than or equal to 500 ms, using Bazett's formula, unless written permission to enroll is provided by the investigator after consultation with a pediatric cardiologist.
* Participant has a clinically significant ECG abnormality (eg, unstable arrhythmia) during screening that, in the opinion of the investigator, could pose a risk to participant safety or interfere with the trial evaluation.
* Within the 3 Months Prior to Screening:
* New onset or worsening of a pre-existing seizure disorder.
* Participants on anti-convulsant medication must be on a stable and therapeutic dose for 3 months prior to screening (if blood level monitoring is clinically available, then the participant must have a therapeutic blood level within 1 week of enrollment).

Other Exclusions:

* Female participant is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 3 months after the last dose of etelcalcetide. (Females of childbearing potential should only be included in the trial after a confirmed menstrual period and a negative highly sensitive serum pregnancy test within 7 days prior to the first dose of investigational product).
* Female participants of childbearing potential unwilling to use 1 highly effective or acceptable method of effective contraception during treatment and for an additional 3 months after the last dose of investigational product.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening by a serum pregnancy test.
* Participant has known sensitivity to etelcalcetide or excipients to be administered during dosing.
* Participant likely to not be available to complete all protocol-required trial visits or procedures, and/or to comply with all required trial procedures to the best of the participant and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) or unacceptable physical findings, that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the trial evaluation procedures or completion.
* Participant has previously entered this trial or previously received treatment with etelcalcetide (Original protocol, Amendment 1 and Amendment 2 only).
* Participant previously has entered this trial (Amendment 3 and later only).
* Anemia, which in the opinion of the investigator makes it not advisable to undergo sequential blood draws.
* History of unstable chronic heart failure within the last 1 year prior to screening.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in iPTH at Weeks 20 to 26 | Week 20 to 26
  To evaluate the efficacy of etelcalcetide in reducing the iPTH level in children ages equal to or greater than 2 to less than 18 years with SHPT receiving maintenance hemodialysis.

SECONDARY OUTCOMES:
Number of Participants Who Achieve a >30% Reduction From Baseline in Mean iPTH | Week 20 to 26
  To evaluate the efficacy of etelcalcetide.
Percent Change From Baseline in Corrected Total Serum Ca and Serum Phosphorus | Week 20 to 26
  To characterize change in laboratory markers of chronic kidney disease.
Proportion of Participants Achieving Corrected Serum Ca Levels Less Than 8.0 mg/dL (2.0 mmol/L) | During the treatment period (up to 31 weeks)
  To characterize the safety of etelcalcetide treatment based on laboratory values.
Proportion of Participants with Hypocalcemia | During the treatment period (up to 31 weeks)
  To characterize the safety of etelcalcetide treatment based on laboratory values.
  Hypocalcemia is defined as corrected serum calcium levels less than 8.4 mg/dL.
Etelcalcetide Plasma Concentrations Before and at the end of Dialysis After Single and Multiple Doses | During the treatment period (up to 31 weeks)
  Etelcalcetide plasma concentrations before and at the end of dialysis after single and multiple doses.
Maximum-observed Concentration (Cmax) of Etelcalcetide | During the treatment period (up to 31 weeks)
  Etelcalcetide plasma concentrations before and at the end of dialysis after single and multiple doses.
Plasma Trough Concentrations (Cmin) of Etelcalcetide | During the treatment period (up to 31 weeks)
  To characterize the PK of etelcalcetide treatment after single and multiple doses.
Number of Participants who Experienced Treatment-emergent Adverse Events (TEAEs) | During the treatment period (up to 31 weeks)
  To characterize the safety of etelcalcetide treatment based on adverse events. Nature, frequency, severity, and relationship to treatment of all adverse events, including those of special interest reported during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Fakultni nemocnice v Motole, Prague, Czechia
- France (2):
  - Hospices Civils de Lyon Hopital Femme Mere Enfant, Bron
  - Hopital Armand Trousseau, Paris
- Germany (5):
  - Kindernierenzentrum Bonn, Bonn
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Zentrum fuer Kinder und Jugendmedizin, Heidelberg
- Greece (2):
  - General Children Hospital Panagioti and Aglaias Kyriakou, Athens
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Azienda Ospedaliera Universitaria Meyer, Florence, Italy
- Childrens Hospital, Affiliate of Vilnius University Hospital Santaros Klinikos, Vilinus, Lithuania
- Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow, Poland
- Unidade Local de Saude de Santo Antonio, EPE - Hospital de Santo Antonio, Porto, Portugal
- Spain (2):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
- United Kingdom (4):
  - Royal Hospital for Sick Children, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Great Ormond Street Hospital for Children, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities.There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com